CLINICAL TRIAL: NCT02029638
Title: Bone Marrow Transplantation and High Dose Post-Transplant Cyclophosphamide for Chimerism Induction and Renal Allograft Tolerance (ITN054ST)
Brief Title: BMT and High Dose Post-Transplant Cyclophosphamide for Chimerism Induction and Renal Allograft Tolerance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN054ST; ACCEPTOR (Other: Immune Tolerance Network (ITN))
Record Dates: First submitted 2013-12-30; First posted 2014-01-08 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Kidney Transplantation
Keywords: renal transplantation; conditioning regimen; BMT; high dose post-transplant cyclophosphamide (PT/Cy); renal allograft tolerance; immunosuppression withdrawal
MeSH Terms: interventions — Antilymphocyte Serum; thymoglobulin; fludarabine; Cyclophosphamide; Whole-Body Irradiation; Acetaminophen; Diphenhydramine; Methylprednisolone; Bone Marrow Transplantation; Mesna; Mycophenolic Acid; Prednisone; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RICG, BMT and high dose PT/Cy+SOC (Experimental): Reduced-intensity conditioning regimen (RICG), bone marrow transplantation (BMT), high dose post-transplant cyclophosphamide (PT/Cy) and Standard of Care (SOC).
  Participants will receive: ATG (pre-transplant), pre-medicated with acetaminophen, diphenhydramine; steroid taper of methylprednisolone; fludarabine (2-6 days before transplant), and low-dose cyclophosphamide (pre- transplant); total body irradiation the day before transplant. Participants will receive a living renal transplant followed by BMT. High-dose cyclophosphamide will be given on days 3 and 4 post-transplant with MESNA. Filgrastim will be given on day 5 post-transplant and continue until absolute neutrophil recovery. Standard immunosuppression of tacrolimus, MMF, and prednisone will begin on day 5 post-transplant and be given ≥26 weeks post-transplant. Eligible participants will be gradually withdrawn from medication over a period of 24-40 weeks.
  Interventions: Biological: anti-thymocyte globulin; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Drug: acetaminophen; Drug: diphenhydramine; Drug: methylprednisolone; Biological: bone marrow transplant; Drug: MESNA; Drug: mycophenolate mofetil; Drug: prednisone; Drug: filgrastim

INTERVENTIONS:
Biological: anti-thymocyte globulin — An initial dose of 0.5 mg/kg IV will be administered over 6 hours on Day -9. Thereafter the daily dose will be increased to 2 mg/kg IV given over 4 hours on Days -8 and -7. No more than 150 mg of ATG may be administered per day.
  Other Names: ATG; Thymoglobulin
Drug: Fludarabine — Fludarabine at dose 30 mg/m^2 will be administered daily by intravenous infusion over 30 minutes on Day -6 to Day -2.
Drug: Cyclophosphamide — 1. Low dose pre-transplant cyclophosphamide will be administered intravenously (IV) over 1- 2 hours, (depending on volume) on Days -6 and -5. The dose of pre-transplant cyclophosphamide is 14.5 mg/kg/day.
  2. High dose cyclophosphamide [50mg/kg (Ideal Body Weight)] will be administered on Day 3 post-transplant (within 60 to 72 hours of marrow infusion) and on Day 4 post-transplant. Cyclophosphamide will be given IV over 1-2 hours depending on volume.
  Other Names: cytoxan
Radiation: Total Body Irradiation — Total body irradiation, consisting of 200 centigray (cGy) Anterior-Posterior/Posterior-Anterior (AP/PA) with 4 Megavolts (MV) or 6 MV photons at 8-12 cGy/min at the point of prescription will be administered in a single day on Day -1.
  Other Names: TBI
Drug: acetaminophen — 650 mg orally prior to antithymocyte globulin infusion.
  Other Names: Tylenol
Drug: diphenhydramine — 25mg diphenhydramine orally prior to antithymocyte globulin infusion.
  Other Names: benadryl
Drug: methylprednisolone — On Days -9 to -7 methylprednisolone 1mg/kg IV 1 hour prior ATG. This dose may be repeated once 3 hours after the first dose of steroids. On Day -6 and -5, methylprednisolone 0.75 mg/kg/ IV as a single dose; on Days -4 and -3, methylprednisolone 0.5 mg/kg/ IV as a single dose; on Day -2 methylprednisolone 0.25 mg/kg/ IV as a single dose.
Biological: bone marrow transplant — Unprocessed, unmanipulated bone marrow will be harvested from the donor and infused into the recipient on Day 0.
  Other Names: bone marrow transfusion; BMT
Drug: MESNA — A series of MESNA doses will be administered for each dose of high dose, post-transplant cyclophosphamide. The total daily dose of MESNA is equal to 80% of the total daily dose of cyclophosphamide.
  Other Names: Mesnex
Drug: mycophenolate mofetil — MMF will be administered at a dose of 15 mg/kg orally three times per day based upon actual body weight, with the maximum of 3 grams a day from Day 5 to 35. The dose will then be reduced to the standard 1 g twice daily thereafter.
  Other Names: MMF; CellCept
Drug: prednisone — Prednisone will be administered at a dose of 10 mg orally daily from Day 5 for 12 weeks. Thereafter the dose will be reduced to 5 mg orally daily.
Drug: filgrastim — All recipients will receive 5 microgram/kg per day of filgrastim as a single, subcutaneous injection from Day 5 post-transplant until the absolute neutrophil count is greater than 1000/µl on three consecutive measurements over at least 2 days.
  Other Names: neupogen

SUMMARY:
The primary objective of this study is to assess the ability of bone marrow transplantation (BMT) and high-dose post-transplantation cyclophosphamide (PT/Cy) to induce renal allograft tolerance and thus enable discontinuation of immunosuppressive therapy in haploidentical living related donor renal transplant recipients.

DETAILED DESCRIPTION:
Transplantation is a good treatment for people with end-stage kidney disease. However, there is still much to learn about how to best care for the transplanted kidney and keep it working for a long time. Unless a person receiving a kidney from someone else takes drugs that reduce immune function, the kidney will be rejected. Those drugs must be continued life-long and cause many issues. Therefore, tolerance of the transplanted kidney, without chronic rejection and without the need for permanent immunosuppressive drug treatment, is a highly desirable goal. If this can be achieved, it would make "one kidney for life" possible.

The study treatment includes several days of study medications followed by a kidney and bone marrow transplant. After the transplant, the study treatment will continue with a few more doses of study medications and then anti-rejection medication is started. After a while, the anti-rejection medication is slowly stopped. Researchers will examine blood and tissue samples and try to identify genetic markers for certain conditions like chimerism, response to therapy, and tolerance.

*** IMPORTANT NOTICE: *** The National Institute of Allergy and Infectious Diseases and the Immune Tolerance Network do not recommend the discontinuation of immunosuppressive therapy for recipients of cell, organ, or tissue transplants outside of physician-directed, controlled clinical studies. Discontinuation of prescribed immunosuppressive therapy can result in serious health consequences and should only be performed in certain rare circumstances, upon the recommendation and with the guidance of your health care provider.

ELIGIBILITY:
Inclusion Criteria:

* Recipient participants must meet all of the following criteria to be eligible for this study:

  * Recipient of a first renal allograft from an Human Leukocyte Antigen (HLA)-haploidentical, living related donor. The donor and recipient must be HLA identical for at least one allele (using high resolution DNA based typing) at the following genetic loci: HLA-A, HLA-B, HLA-C and HLA-DRB1. Fulfillment of this criterion shall be considered sufficient evidence that the donor and recipient share one HLA haplotype.
  * Age 18 to 65 years.
  * Single solid organ recipients (kidney only).
  * Blood Group System (ABO) compatibility with donor.
  * Donor-Specific Antibody (DSA) will be assessed by the local laboratory 30 days or less prior to transplant using solid phase micro particle technology (by Luminex® phenotype panel or Luminex single antigen bead test.) The following criteria apply:
* Participants without detectable DSA will be deemed eligible if they meet other entry criteria.
* Participants with detectable DSA and a positive flow cytometric crossmatch may undergo de-sensitization per standard of care if they are cytotoxic crossmatch negative. Such participants must demonstrate a negative flow cytometric crossmatch by day -9 in order to receive the first dose of study therapy (ATG). Participants who do not demonstrate an acceptable response to de-sensitization by day -9 will be considered screen failures and will be terminated from the study.
* Participants with a positive cytotoxicity crossmatch will be excluded.
* No known history of anti-HLA antibodies. Recipients with low- level anti-HLA antibodies not considered to be clinically significant may be eligible, following consultation with the Protocol Chairs, the local HLA Laboratory Director, the NIAID Medical Monitor and the ITN Clinical Trial Physician.
* Negative T and B cell flow crossmatches with the designated donor; as assessed by local laboratories. If one or more of the crossmatches is positive, the participant will be considered a screen failure unless combined results of antibody and cross match testing implicate a non-HLA antibody as the cause of the positive flow crossmatch. In this case, the Protocol Chair must approve the participant as a screening success after consultation with the local HLA Laboratory Director.
* Normal estimated left ventricular ejection fraction and no history of ischemic heart disease requiring revascularization, unless cleared by a cardiologist.
* Forced expiratory volume (FEV1) and forced vital capacity (FVC) > 40% of predicted at the screening visit.
* Serological evidence of prior Epstein-Barr virus (EBV) infection as documented by positive IgG and negative IgM antibodies against EBV.
* For women of childbearing potential, a negative serum or urine pregnancy test with sensitivity less than 50 Milli-International unit (mIU)/m within 72 hours before the start of study medication.
* Use of two forms of contraception with less than a 5% failure rate or abstinence by all transplanted participants for 18 months after the first dose of study therapy. For the first 60 days post-transplant, recipients should be encouraged to use non-hormonal contraceptives due to the potential adverse effect of hormones on bone marrow engraftment.
* Ability to receive oral medication.
* Ability to understand and provide informed consent.
* All participants must demonstrate a negative QuantiFERON® (QFT) assay result within 52 weeks of transplant regardless of Purified Protein Derivative (PPD) status. Participants with a positive QFT assay will not be eligible for the study unless they have completed treatment for latent TB and have a negative chest x-ray. QFT testing done within 52 weeks before transplant is acceptable as long as there is documentation of the results. Prior recipients of a Bacillus Calmette-Guérin (BCG) vaccination are not exempt.
* Donor participants must meet all of the following criteria to be eligible for this study:

  * HLA-haploidentical, first-degree relatives or half-siblings of the recipient participant at the allele or allele group. The donor and recipient must be HLA identical for at least one allele (using high resolution DNA based typing) at the following genetic loci: HLA-A, HLA-B, HLA-C, and HLA-DRB1. Fulfillment of this criterion shall be considered sufficient evidence that the donor and recipient share one HLA haplotype.
  * Age 18 to 65 years.
  * Creatinine clearance >80 ml/minute as measured from a 24 hour urine collection within 26 weeks of the screening visit. If a serum creatinine drawn at the screening visit is > 20% higher than the serum creatinine drawn at the time of the 24 urine collection, the creatinine clearance must be re-evaluated by a repeat 24 hour urine test. If the new value is ≤80mg/dL the donor will be excluded.
  * Meets institutional selection criteria for organ and bone marrow donation.
  * Ability to understand and provide informed consent for all study procedures including kidney transplant and bone marrow harvest.
  * Serologic evidence of prior EBV infection as documented by positive Immunoglobulin G (IgG) and negative Immunoglobulin M (IgM) antibodies against EBV.

Exclusion Criteria:

* Recipient subjects who meet any of the following criteria will not be eligible for this study:

  * Underlying renal disease with a high risk of disease recurrence in the transplanted kidney, including:

    1. Focal segmental glomerulosclerosis (FSGS).
    2. Type I or II membranoproliferative glomerulonephritis.
    3. Hemolytic-uremic syndrome/thrombotic thrombocytopenic purpura.
  * Clinically important genital/urinary tract dysfunction.
  * Body mass index (BMI) > 40.
  * Women who are breastfeeding.
  * History of cancer within the last 5 years, except for nonmelanoma skin cancer, stage 1 renal cell carcinoma, stage 1 prostate cancers cured by local resection and any curatively treated carcinomas in situ.
  * History of positive HIV-1 or HIV-2 serologies or nucleic acid test.
  * Evidence of prior hepatitis B infection as evaluated by hepatitis B surface antigen (HBsAg), total hepatitis B core antibody (anti-HBc IgM and IgG) and Hepatitis B surface antibody (anti-HBsAb).

Subjects demonstrating any one of the following will be excluded:

* Positive hepatitis B surface antigen (HBsAg) or
* Positive anti-HBc IgM.
* Positive anti-HBc IgG.
* Positive Hepatitis B virus (HBV) Polymerase chain reaction (PCR).
* Positive anti-hepatitis C (HCV) antibodies and a positive serum HCV RNA PCR. All positive HCV antibody results must be assessed by an Electroimmunoassay (EIA) assay and confirmed by a quantitative serum HCV RNA assay. Participants with positive HCV antibodies but undetectable serum HCV RNA may be considered for eligibility. Participants with negative anti-HCV antibodies but unexplained liver enzyme abnormalities must undergo a quantitative serum RNA assay to rule out false negative HCV serologies.
* History of active Tuberculosis (TB).
* Any active, severe local or systemic infection at the screening visit.
* Autoimmune disease requiring immunosuppressive drugs for maintenance.
* Use of investigational drug, other than the study medications specified by the protocol, within 30 days of transplantation.
* Receipt of a live vaccine within 30 days of receipt of study therapy.
* The presence of any medical condition that the Investigator deems incompatible with participation in the trial.
* Donor subjects who meet any of the following criteria will not be eligible for this study:

  * History of type I or type II diabetes mellitus.
  * History of severe cardiovascular disease, defined as New York Heart Association Class III or IV.
  * History of blood product donation to recipient.
  * History of positive HIV-1 or HIV-2 serology or nucleic acid test.
  * Evidence of prior hepatitis B infection.

Subjects demonstrating any one of the following will be excluded:

* Positive hepatitis B surface antigen (HBsAg) or
* Positive anti- hepatitis B core antigen (HBc) IgM.
* Positive anti-HBc IgG.
* Positive HBV PCR
* Positive anti-hepatitis C (HCV) antibodies and a positive serum HCV RNA PCR. All positive HCV antibody results must be assessed by an EIA assay and confirmed by a quantitative serum HCV RNA assay. Participants with positive HCV antibodies but undetectable serum HCV RNA may be considered for eligibility. Participants with negative anti-HCV antibodies but unexplained liver enzyme abnormalities must undergo a quantitative serum RNA assay to rule out false negative HCV serologies.
* Autoimmune disease requiring immunosuppressive drugs for maintenance.
* The presence of any medical condition that the Investigator deems incompatible with participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lode Swinnen, MD, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Solez K, Colvin RB, Racusen LC, Haas M, Sis B, Mengel M, Halloran PF, Baldwin W, Banfi G, Collins AB, Cosio F, David DS, Drachenberg C, Einecke G, Fogo AB, Gibson IW, Glotz D, Iskandar SS, Kraus E, Lerut E, Mannon RB, Mihatsch M, Nankivell BJ, Nickeleit V, Papadimitriou JC, Randhawa P, Regele H, Renaudin K, Roberts I, Seron D, Smith RN, Valente M. Banff 07 classification of renal allograft pathology: updates and future directions. Am J Transplant. 2008 Apr;8(4):753-60. doi: 10.1111/j.1600-6143.2008.02159.x. Epub 2008 Feb 19. PMID 18294345
- See also: National Institute of Allergy and Infectious Diseases website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled, Screen Failure: Participants were consented and enrolled in the study, but did not receive a full evaluation of all criteria for study participation. These participants were terminated during the screening process due to a decision by study sponsor
- Enrolled, Not Transplanted: Participants were consented and enrolled in the study, fulfilling all criteria for study participation. The participants initiated protocol specified pre-transplant treatment, but did not receive a renal transplantation followed by bone marrow infusion, per protocol.
- Enrolled, Transplanted: Participants were consented, enrolled, fulfilling all study criteria. Participants received three .5, 2, and 2 mg/kg doses of ATG (7-9 days before transplant) pre-medicated with 650 mg acetaminophen, 25 mg diphenhydramine and steroid taper of methylprednisolone, five 30 mg/m^2/day doses of fludarabine (2-6 days before transplant), and two 14.5 mg/kg/day doses of low-dose cyclophosphamide (5-6 days before transplant), along with total body irradiation the day before transplant. Participants received a living renal transplant followed by bone marrow infusion. Two 50 mg/kg/day doses of high-dose cyclophosphamide were given days 3 and 4 post-transplant with MESNA. Filgrastim was given starting on day 5 post-transplant until absolute neutrophil recovery. Standard immunosuppression of tacrolimus, MMF, and prednisone began on day 5 post-transplant and given for at least 26 weeks post-transplant. Eligible participants were gradually withdrawn from medication over a period of 24-40 weeks.
Period: Overall Study
Arm/Group | Enrolled, Screen Failure | Enrolled, Not Transplanted | Enrolled, Transplanted
Started | 2 | 1 | 1
Completed | 0 | 1 | 0
Not Completed | 2 | 0 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Decision by Study Sponsor or Regulatory | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Enrolled, Screen Failure | Enrolled, Not Transplanted | Enrolled, Transplanted | Total
Number analyzed (Participants) | 2 | 1 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 1 | 4
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 1 | 0 | 1 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 1 | 4
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] — Serum creatinine (Cr) is an indicator of kidney function. Cr is a substance formed from the metabolism of creatine, commonly found in blood, urine, and muscle tissue. It is removed from the blood by the kidneys and excreted in urine.The baseline Cr interval per protocol is defined as the interval prior to immunosuppressive maintenance withdrawal (IMW) initiation.This is the 2 to 4 week interval post-kidney transplant, calculated using the lowest 3 serum Cr values during this pre-defined interval (excluded:days on dialysis). Normal:adult males, 0.7 to 1.3 mg/dL; adult females, 0.6 to 1.1 mg/dL.
  mg/dL | NA (NA) — Participants in this group did not have data to contribute to this baseline measure since they did not receive a transplant. | NA (NA) — Participants in this group did not have data to contribute to this baseline measure since they did not receive a transplant. | 2.1 (NA) — Standard deviation cannot be calculated for one participant. | 2.1 (NA) — Standard deviation cannot be calculated for one participant.

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Achieved Operational Tolerance
Description: Operational tolerance is defined as remaining off all immunosuppression 52 weeks after completion of immunosuppression withdrawal, with no evidence of biopsy-proven allograft rejection and, with acceptable renal function defined as a serum creatinine that has increased no more than 25% above baseline at the primary endpoint visit. Baseline creatinine is defined as the average of the lowest three creatinine values during 2 to 4 weeks post-transplant, excluding days on dialysis. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through 52 Weeks after Discontinuation of All Immunosuppression
Population: Transplanted Per Protocol Participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Enrolled, Transplanted: Participants were consented, enrolled, and fulfilled all study criteria. Participants received three .5, 2, and 2 mg/kg doses of ATG (7-9 days before transplant) pre-medicated with 650 mg acetaminophen, 25 mg diphenhydramine and steroid taper of methylprednisolone, five 30 mg/m^2/day doses of fludarabine (2-6 days before transplant), and two 14.5 mg/kg/day doses of low-dose cyclophosphamide (5-6 days before transplant), along with total body irradiation the day before transplant. Participants received a living renal transplant followed by bone marrow infusion. Two 50 mg/kg/day doses of high-dose cyclophosphamide were given days 3 and 4 post-transplant with MESNA. Filgrastim was given starting on day 5 post-transplant until absolute neutrophil recovery. Standard immunosuppression of tacrolimus, MMF, and prednisone began on day 5 post-transplant and given for at least 26 weeks post-transplant. Eligible participants were gradually withdrawn from medication over a period of 24-40 weeks.
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Percent of participants | 0 [0 to 97.5]

2. Secondary Outcome: Number of Participants Experiencing an Incidence of Graft-versus-Host Disease Post-Transplant
Description: Graft-versus-host disease (GVHD) is a medical complication that can occur after a person receives transplanted tissue, most commonly occurring after a bone marrow transplant. The white blood cells from the donated tissue recognize the tissue recipient's cells as foreign. These donor cells then attack the recipient's cells.
Time Frame: Transplant to Two Years Post-Transplant
Population: Transplanted Per Protocol Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Severity of Graft-versus-Host Disease in Transplanted Participants
Description: Graft-versus-host disease (GVHD) is a medical complication that can occur after a person receives transplanted tissue, most commonly occurring after a bone marrow transplant. The white blood cells from the donated tissue recognize the tissue recipient's cells as foreign. These donor cells then attack the recipient's cells. Severity of GVHD is based on skin, liver, and intestinal tract symptoms, ranging from I to IV, with IV being the worst. This measure counts the number of participants experiencing GVHD by severity.
Time Frame: Transplant to Two Years Post-Transplant
Population: Transplanted Per Protocol Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Participants
  Grade I | 1
  Grade II | 0
  Grade III | 0
  Grade IV | 0

4. Secondary Outcome: Duration in Days of Graft-versus-Host Disease in Transplanted Participants
Description: Graft-versus-host disease (GVHD) is a medical complication that can occur after a person receives transplanted tissue, most commonly occurring after a bone marrow transplant. The white blood cells from the donated tissue recognize the tissue recipient's cells as foreign. These donor cells then attack the recipient's cells. Duration (in days) is measured as the time from the start of the GVHD event to the end of the GVHD event.
Time Frame: Transplant to Two Years Post-Transplant
Population: Transplanted Per Protocol Participants
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Enrolled, Transplanted: .Participants were consented, enrolled, and fulfilled all study criteria. Participants received three .5, 2, and 2 mg/kg doses of ATG (7-9 days before transplant) pre-medicated with 650 mg acetaminophen, 25 mg diphenhydramine and steroid taper of methylprednisolone, five 30 mg/m^2/day doses of fludarabine (2-6 days before transplant), and two 14.5 mg/kg/day doses of low-dose cyclophosphamide (5-6 days before transplant), along with total body irradiation the day before transplant. Participants received a living renal transplant followed by bone marrow infusion. Two 50 mg/kg/day doses of high-dose cyclophosphamide were given days 3 and 4 post-transplant with MESNA. Filgrastim was given starting on day 5 post-transplant until absolute neutrophil recovery. Standard immunosuppression of tacrolimus, MMF, and prednisone began on day 5 post-transplant and given for at least 26 weeks post-transplant. Eligible participants were gradually withdrawn from medication over a period of 24-40 weeks.
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Days | 7 (NA) — Standard deviation cannot be calculated for one participant.

5. Secondary Outcome: Number of Transplanted Participants With Engraftment Syndrome
Description: Engraftment syndrome is a complication that can occur following bone marrow transplant. The presence of engraftment syndrome is diagnosed by monitoring the common symptoms, which include: fever, rash, fluid in the lungs, and serum creatinine values above 4 mg/dL occurring within a week of absolute neutrophil recovery (e.g., first day after three consecutive daily absolute neutrophil counts ≥ 500 per µL), without apparent other cause.
Time Frame: Transplant to End of Study (Up to 25 months After Enrollment)
Population: Transplanted Per Protocol Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Duration in Days of Engraftment Syndrome in Transplanted Participants
Description: Engraftment syndrome is a complication that can occur following bone marrow transplant. The presence of engraftment syndrome is diagnosed by monitoring the common symptoms, which include: fever, rash, fluid in the lungs, and serum creatinine values above 4 mg/dL occurring within a week of absolute neutrophil recovery (e.g., first day after three consecutive daily absolute neutrophil count ≥ 500 per µL), without apparent other cause. Duration (in days) is measured as the time from the start of the engraftment syndrome event to the end of the engraftment syndrome event.
Time Frame: Transplant to End of Study (Up to 25 months After Enrollment)
Population: No statistical analyses provided for 'Duration of Engraftment Syndrome in Transplanted Participants' because no participants in the Per Protocol population experienced engraftment syndrome.
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Transplanted Participants Who Died
Description: Number of participant deaths after receiving a transplant per protocol.
Time Frame: Transplant to End of Study (Up to 25 months After Enrollment)
Population: Transplanted Per Protocol Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Participants | 1

8. Secondary Outcome: Number of Transplanted Participants With Acute Renal Allograft Rejection
Description: Acute renal allograft rejection demonstrated either by biopsy or clinically (when a biopsy could not be performed). This measure includes participants with biopsy proven acute renal allograft rejection and those that have creatinine values 25% or greater relative to baseline for over 72 hours. Baseline serum creatinine is defined as the average of the lowest three serum creatinine values during 2 to 4 weeks post-transplant, excluding days on dialysis.
Time Frame: Transplant to End of Study (Up to 25 months After Enrollment)
Population: Transplanted Per Protocol Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Participants | 1

9. Secondary Outcome: Histological Severity of Biopsies Demonstrating Acute Rejection as Defined by Banff 2007 Classification Renal Allograft Pathology
Description: This outcome includes results from biopsies with proven acute renal allograft rejection according to the 2007 Banff Classification Renal Allograft Pathology. A Banff result of indeterminate is not classified as rejection.
Time Frame: Transplant to End of Study (Up to 25 months After Enrollment)
Population: Transplanted Per Protocol Participants
Measure: Number; unit: participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
participants
  Acute Cellular Rejection Banff Grade IA | 0
  Acute Cellular Rejection Banff Grade IB | 0
  Acute Cellular Rejection Banff Grade IIA | 0
  Acute Cellular Rejection Banff Grade IIB | 0
  Acute Cellular Rejection Banff Grade III | 0
  Acute Antibody Mediated Rejection | 0

10. Secondary Outcome: Number of Transplanted Participants With Chronic T Cell-Mediated or Antibody-Mediated Rejection
Description: Outcome includes participants who experienced chronic T cell-mediated rejection, antibody-mediated rejection and progressive interstitial fibrosis/tubular atrophy (IF/TA), transplant glomerulopathy or chronic obliterative arteriopathy, without an alternative, non-rejection related cause. Reference: Banff 2007 Classification Renal Allograft Pathology definition of terms.
Time Frame: Transplant to End of Study (Up to 25 months After Enrollment)
Population: Transplanted Per Protocol Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Participants | 1

11. Secondary Outcome: Number of Days Post-Transplant to the First Episode of Acute Rejection Requiring Treatment
Description: Number of days post-transplant to the first episode of acute rejection that required treatment. This includes acute rejection episodes requiring treatment that were not biopsy proven.
Time Frame: Transplant to End of Study (Up to 25 months After Enrollment)
Population: Transplanted Per Protocol Participants who experienced acute rejection.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Days | 23 (NA) — Standard deviation cannot be calculated for one participant.

12. Secondary Outcome: Number of Adverse Events (AEs)- Including Infection, Wound Complications, Post-transplant Diabetes, Hemorrhagic Cystitis and Malignancy
Description: AEs reported as an infection, wound complication, post-transplant diabetes, hemorrhagic cystitis and/or malignancy.
Time Frame: First Dose of Study Medication to End of Study (Up to 25 Months After Enrollment)
Population: Safety population, which includes all participants who received any study medication.
Measure: Number; unit: Events
Groups:
- Enrolled, Not Transplanted: Participants were consented and enrolled in the study, but did not receive a full evaluation of all criteria for study participation. These participants were terminated during the screening process due to a decision by study sponsor.
Arm/Group | Enrolled, Not Transplanted | Enrolled, Transplanted
Number analyzed (Participants) | 1 | 1
Events
  Infection | 0 | 2
  Wound complications | 0 | 0
  Post-transplant diabetes | 0 | 0
  Hemorrhagic cystitis | 0 | 0
  Malignancy | 0 | 0

13. Secondary Outcome: Number of Adverse Events (AEs) by Severity- Including Infection, Wound Complications, Post-Transplant Diabetes, Hemorrhagic Cystitis and Malignancy
Description: AEs reported as an infection, wound complication, post-transplant diabetes, hemorrhagic cystitis and/or malignancy. Grades are based on National Cancer Institute--Common Terminology Criteria (NCI-CTCAE) Version 4.0.
Time Frame: First Dose of Study Medication to End of Study (Up to 25 Months After Enrollment)
Population: Safety population, which includes all participants who received any study medication.
Measure: Number; unit: Events
Arm/Group | Enrolled, Not Transplanted | Enrolled, Transplanted
Number analyzed (Participants) | 1 | 1
Events
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 2
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

14. Secondary Outcome: Duration in Days of Adverse Events (AEs)- Including Infection, Wound Complications, Post-transplant Diabetes, Hemorrhagic Cystitis and Malignancy
Description: AEs reported as an infection, wound complication, post-transplant diabetes, hemorrhagic cystitis and/or malignancy. Time (in days) from the start date of the AE until the end date of the AE. Two events contributed to this calculation.
Time Frame: First Dose of Study Medication to End of Study (Up to 25 Months After Enrollment)
Population: Participants who received any study medication and experienced at least one AE inclusive of infection, wound complications, post-transplant diabetes, hemorrhagic cystitis and/or malignancy.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enrolled, Not Transplanted | Enrolled, Transplanted
Number analyzed (Participants) | 0 | 1
Days |  | 9.5 (2.12)

15. Secondary Outcome: Number of Transplanted Participants Who Developed Donor- Specific Antibody After Initiation of Immunosuppression Withdrawal
Description: Donor-specific antibodies are directed against antigens expressed on donor organs. These antibodies can result in an immune attack on the transplanted organ, increasing risk of graft loss and/or rejection.
Time Frame: Initiation of Immunosuppression Withdrawal to End of Study (to 25 months)
Population: Transplanted Per Protocol Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Participants | 0

16. Secondary Outcome: Number of Transplanted Participants Who Developed Donor-Specific Antibody During Study Participation
Description: as for outcome 15
Time Frame: Transplant to End of Study (Up to 25 months)
Population: Transplanted Per Protocol Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Participants | 0

17. Secondary Outcome: Number of Days From Neutrophil Nadir to Absolute Neutrophil Recovery
Description: Time (in days) from neutrophil nadir, the first day post-transplant on which the absolute neutrophil count (ANC) is below 500 per µL, to the first day after three consecutive daily ANCs ≥ 500 per µL. ANC is a measure of the number of neutrophils present in the blood. Neutrophils are a type of white blood cell that fight against infection. A healthy person has an ANC between 2,500 and 6,000 per µL. A value below 500 per µL means the risk of infection is higher.
Time Frame: Post-Transplant Neutrophil Nadir to Neutrophil Recover
Population: Transplanted Per Protocol Participants
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Days | 15 (NA) — Standard deviation cannot be calculated for one participant.

18. Secondary Outcome: Number of Days From Transplant to Platelet Count Recovery
Description: Time (in days) from transplant to the first day of a platelet count of ≥20,000 per μL without a prior platelet transfusion in the preceding seven days. Low platelet numbers is associated with increased risk of bleeding and bruising. A healthy person has a platelet count ranging from 150,000 to 450,000 platelets per microliter of blood.
Time Frame: Transplant to Platelet Count Recovery
Population: Transplanted Per Protocol Participants
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Days | 36 (NA) — Standard deviation cannot be calculated for one participant.

19. Secondary Outcome: Number of Transplanted Participants Who Remained Off Immunosuppression for at Least 52 Weeks, Including Those in Whom the 52 Week Biopsy Was Not Performed
Description: Number of transplanted participants who remained off immunosuppression for ≥52 weeks, including those in whom the 52 week biopsy was not performed. This outcome included participants who were able to withdrawal successfully from all immunosuppression medication and remain off all immunosuppression for 52 weeks after the completion of withdrawal.
Time Frame: Transplant to 52 Weeks after Discontinuation of All Immunosuppression
Population: Transplanted Per Protocol Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Participants | 0

20. Secondary Outcome: Number of Participants Free From Return to Immunosuppression for the Duration of the Study
Description: Participants who were able to withdrawal successfully from all immunosuppression medication and remained off all immunosuppression medication for the remainder of the study.
Time Frame: Transplant to End of Study (Up to 25 Months)
Population: Transplanted Per Protocol Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled, Transplanted
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: First study medication dosing through end of study (up to 25 months after enrollment)
Arm/Group | Enrolled, Not Transplanted | Enrolled, Transplanted
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled, Not Transplanted (N=1) | Enrolled, Transplanted (N=1)
Benign intracranial hypertension (Nervous system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled, Not Transplanted (N=1) | Enrolled, Transplanted (N=1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Acute graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to slow accrual and a current assessment of risks related to the study, the study was closed to enrollment in December 2016. Participants actively screening did not move forward in the study and those on trial completed safety follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT02029638/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT02029638/SAP_001.pdf